CLINICAL TRIAL: NCT00044213
Title: Trial to Assess Chelation Therapy (TACT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mt. Sinai Medical Center, Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gervasio Lamas, MD, Chair, Department of Medicine- Chief, Division of Cardiology, Mt. Sinai Medical Center, Miami
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 654; U01HL092607 (NIH); U01AT001156 (NIH)
Record Dates: First submitted 2002-08-22; First posted 2002-08-23 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Edetic Acid; Vitamins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EDTA + high dose vitamin (Active Comparator): Participants will receive 40 infusions of active EDTA chelation and active high-dose oral vitamins.
  Interventions: Drug: EDTA; Dietary Supplement: High Dose Vitamin
- EDTA + high dose vitamin placebo (Placebo Comparator): Participants will receive 40 infusions of EDTA chelation and placebo high-dose oral vitamins.
  Interventions: Drug: EDTA; Dietary Supplement: High Dose Vitamin Placebo
- EDTA placebo + high dose vitamin (Placebo Comparator): Participants will receive 40 infusions of placebo EDTA chelation and active high-dose oral vitamins.
  Interventions: Drug: EDTA Placebo; Dietary Supplement: High Dose Vitamin
- EDTA placebo + high dose vitamin placebo (Placebo Comparator): Participants will receive 40 infusions of placebo EDTA chelation and placebo high-dose oral vitamins.
  Interventions: Drug: EDTA Placebo; Dietary Supplement: High Dose Vitamin Placebo

INTERVENTIONS:
Drug: EDTA — Participants will receive 40 infusions of standard chelation solution.
  Arms: EDTA + high dose vitamin; EDTA + high dose vitamin placebo
Drug: EDTA Placebo — Participants will receive 40 infusions of EDTA placebo.
  Arms: EDTA placebo + high dose vitamin; EDTA placebo + high dose vitamin placebo
Dietary Supplement: High Dose Vitamin
  Arms: EDTA + high dose vitamin; EDTA placebo + high dose vitamin
Dietary Supplement: High Dose Vitamin Placebo
  Arms: EDTA + high dose vitamin placebo; EDTA placebo + high dose vitamin placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of ethylene diamine tetra-acetic (EDTA) chelation therapy in individuals with coronary artery disease.

DETAILED DESCRIPTION:
EDTA chelation therapy involves repeated administrations of a synthetic amino acid to reduce atherosclerotic plaque and other mineral deposits throughout the cardiovascular system.

Participants will be randomly assigned to receive 40 infusions of either the standard chelation solution or placebo. The primary endpoint of this trial will be a composite of all cause mortality, myocardial infarction, stroke, coronary revascularization, and hospitalization for angina.

The results of TACT will provide either a significant positive result or an informative null result upon which rational clinical decision-making and health policy can be based.

ELIGIBILITY:
Inclusion Criteria for Participants:

* Heart attack at least 6 weeks prior to study start

Exclusion Criteria for Participants:

* Serum creatinie level greater than 2.0 mg/dL
* Platelet count less than 100,000/µL
* Blood pressure greater than 160/100
* Chelation therapy within 5 years prior to study start
* History of allergic reactions to EDTA or any of the therapy's components
* Coronary or carotid revascularization procedures within 6 months prior to study start or a scheduled revascularization
* Cigarette smoking within 3 months prior to study start
* Childbearing potential
* History of liver disease
* Active heart failure or heart failure hospitalization within 6 months.
* Diagnoses of additional medical conditions that could otherwise limit patient survival
* Inability to tolerate 500-mL infusions weekly.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1708 (Actual)
Dates: Start 2003-09; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gervasio A Lamas, M.D., Study Director — Icahn School of Medicine at Mount Sinai
Locations (86):
- United States (73):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mt Holistic Health Center, Danville, California
  - Patrick A. Golden, Fresno, California
  - Scripps Center for Integrative Medicine, La Jolla, California
  - Phoenix Wellness Group, Napa, California
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - The Blend Institute, Bradenton, Florida
  - Wellness Works, Brandon, Florida
  - Innovative Research of West Florida, Clearwater, Florida
  - Hyperbaric Medicine Inc., Fort Walton Beach, Florida
  - White-Wilson Medical Center, Fort Walton Beach, Florida
  - Tru Med, Melbourne, Florida
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Tri-Health Alternative Medical Center, Mt. Dora, Florida
  - Heart and Vascular Center for Research, Inc., Sarasota, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Life Family Practice Center for Complementary and Alternative Medicine, The Villages, Florida
  - Florida Medical Clinic, P.A. Clinical Research Division, Zephyrhills, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Full Circle Medical Center, Fort Oglethorpe, Georgia
  - Crossroads Healing Arts LLC, Goshen, Indiana
  - Integrative Medical Center at Schneck Medical Center, Seymour, Indiana
  - Northwest Indiana Cardiovascular Physicians Inc., Valparaiso, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - The Center for the Improvement of Functioning International, Wichita, Kansas
  - Complementary Medical Services, Mandeville, Louisiana
  - Maine Integrative Wellness, Portland, Maine
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Marino Center for Progressive Health, Cambridge, Massachusetts
  - Henry Ford Health System Preventative Cardiology Clay Ford Center for Athletic Medicine, Detroit, Michigan
  - The Preventive Medicine Center, Flint, Michigan
  - Born Preventive Health Care Clinic, Grand Rapids, Michigan
  - Parchment Family Practice, Kalamazoo, Michigan
  - Berman Center for Outcomes and Clinical Research, Minneapolis, Minnesota
  - Mayo Clinic and Foundation Cardiovascular Health Clinic, Rochester, Minnesota
  - University of Missouri Hospital and Clinics, Columbia, Missouri
  - Brian Dieterle, MD, PhD, Hollister, Missouri
  - Preventive Medicine, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Magaziner Center for Wellness, Cherry Hill, New Jersey
  - Park Professional Building, Roselle Park, New Jersey
  - Stockton Family Practice, Stockton, New Jersey
  - Heart Care Center, East Syracuse, New York
  - The Gables Natural Medicines Center & Day Spa Family Health Services, Mayville, New York
  - NYU School of Medicine, New York, New York
  - Rhinebeck Health Center, Rhinebeck, New York
  - Staten Island Heart, Staten Island, New York
  - Schachter Center for Complementary Medicine, Suffern, New York
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - Integrative Medical Associates, PLLC, Tryon, North Carolina
  - Celebration of Health Center, Bluffton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Comprehensive Heart Care, Inc., Toledo, Ohio
  - Upper Valley Family Care, Troy, Ohio
  - COR Research, Oklahoma City, Oklahoma
  - St. Charles Health System, Bend, Oregon
  - Center for Environmental Medicine, Portland, Oregon
  - Wholistic Health Center, Greensburg, Pennsylvania
  - Woodlands Healing Research Center, Quakertown, Pennsylvania
  - Main Line Health Heart Center, Wynnewood, Pennsylvania
  - Biogenesis Medical Center, Landrum, South Carolina
  - Athens Surgery Clinic, Athens, Tennessee
  - The Castle Clinic, PLLC, Johnson City, Tennessee
  - Chelation Centers of Texas, Texas City, Texas
  - Freedom Center for Advanced Medicine, Provo, Utah
  - The Cardiovascular Group, Fairfax, Virginia
  - Virginia Beach General Hospital, Virginia Beach, Virginia
  - Hope Medical Holistic Clinic, Vancouver, Washington
  - Care Foundation Inc., Wausau, Wisconsin
  - Waters Preventive Medical Center, LTD, Wisconsin Dells, Wisconsin
- Canada (13):
  - Cline Medical Centre, Nanaimo, British Columbia
  - The Wellness Centre, Port Hawkesbury, Nova Scotia
  - Chelation Center of Barrie, Inc., Barrie, Ontario
  - Anti-Aging & Family Wellness Clinic, Madoc, Ontario
  - Markham Integrative Medicine, Markham, Ontario
  - North Bay Complementary, North Bay, Ontario
  - Seekers Centre for Integrative Medicine, Ottawa, Ontario
  - Dr. C. Minielly, Smith Falls, Ontario
  - Chelation Center of Don Valley Inc., Toronto, Ontario
  - Jaconello Health Centre, Toronto, Ontario
  - Chelation and Natural Therapy, Toronto, Ontario
  - Chelox, Toronto, Ontario
  - Saskatoon Chelation Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Escolar E, Ujueta F, Kim H, Mark DB, Boineau R, Nahin RL, Goertz C, Lee KL, Anstrom KJ, Lamas GA. Possible differential benefits of edetate disodium in post-myocardial infarction patients with diabetes treated with different hypoglycemic strategies in the Trial to Assess Chelation Therapy (TACT). J Diabetes Complications. 2020 Aug;34(8):107616. doi: 10.1016/j.jdiacomp.2020.107616. Epub 2020 May 7. PMID 32446881
- [Derived] Mark DB, Anstrom KJ, Clapp-Channing NE, Knight JD, Boineau R, Goertz C, Rozema TC, Liu DM, Nahin RL, Rosenberg Y, Drisko J, Lee KL, Lamas GA; TACT Investigators. Quality-of-life outcomes with a disodium EDTA chelation regimen for coronary disease: results from the trial to assess chelation therapy randomized trial. Circ Cardiovasc Qual Outcomes. 2014 Jul;7(4):508-16. doi: 10.1161/CIRCOUTCOMES.114.000977. PMID 24987051
- [Derived] Lamas GA, Boineau R, Goertz C, Mark DB, Rosenberg Y, Stylianou M, Rozema T, Nahin RL, Lindblad L, Lewis EF, Drisko J, Lee KL; TACT (Trial to Assess Chelation Therapy) Investigators. Oral high-dose multivitamins and minerals after myocardial infarction: a randomized trial. Ann Intern Med. 2013 Dec 17;159(12):797-805. doi: 10.7326/0003-4819-159-12-201312170-00004. PMID 24490264
- [Derived] Escolar E, Lamas GA, Mark DB, Boineau R, Goertz C, Rosenberg Y, Nahin RL, Ouyang P, Rozema T, Magaziner A, Nahas R, Lewis EF, Lindblad L, Lee KL. The effect of an EDTA-based chelation regimen on patients with diabetes mellitus and prior myocardial infarction in the Trial to Assess Chelation Therapy (TACT). Circ Cardiovasc Qual Outcomes. 2014 Jan;7(1):15-24. doi: 10.1161/CIRCOUTCOMES.113.000663. Epub 2013 Nov 19. PMID 24254885
- [Derived] Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Lindblad L, Lewis EF, Drisko J, Lee KL; TACT Investigators. Effect of disodium EDTA chelation regimen on cardiovascular events in patients with previous myocardial infarction: the TACT randomized trial. JAMA. 2013 Mar 27;309(12):1241-50. doi: 10.1001/jama.2013.2107. PMID 23532240
- [Derived] Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Drisko JA, Lee KL. Design of the Trial to Assess Chelation Therapy (TACT). Am Heart J. 2012 Jan;163(1):7-12. doi: 10.1016/j.ahj.2011.10.002. PMID 22172430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The primary analysis of the trial included 1708 patients who had been enrolled from September 2003 through October 2011 (median, 55 months)Participants were recruited at 134 sites in the US and Canada.
Period: Overall Study
Arm/Group | EDTA + High Dose Vitamin | EDTA + High Dose Vitamin Placebo | EDTA Placebo + High Dose Vitamin | EDTA Placebo + High Dose Vitamin Placebo
Started | 421 | 418 | 432 | 437
Completed | 321 | 306 | 294 | 301
Not Completed | 100 | 112 | 138 | 136
Not completed — Withdrawal by Subject | 50 | 65 | 91 | 83
Not completed — Death | 42 | 42 | 42 | 49
Not completed — Lost to Follow-up | 8 | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EDTA + High Dose Vitamin | EDTA + High Dose Vitamin Placebo | EDTA Placebo + High Dose Vitamin | EDTA Placebo + High Dose Vitamin Placebo | Total
Number analyzed (Participants) | 421 | 418 | 432 | 437 | 1708
Age Continuous [Mean (Full Range); unit: Years] | 65 [59 to 71] | 65 [60 to 72] | 66 [59 to 72] | 66 [59 to 72] | 65.5 [59 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 82 | 77 | 70 | 299
  Male | 351 | 336 | 355 | 367 | 1409

OUTCOME MEASURES:

1. Primary Outcome: A Composite of Total Mortality, Recurrent Myocardial Infarction, Stroke, Coronary Revascularization, and Hospitalization for Angina.
Description: Number of patients with events (composite of death from any cause, MI, stroke, coronary revascularization or hospitalization for angina) Events were centrally adjudicated where available; otherwise site reported events were used.
Time Frame: Measured over a maximum 5-year follow-up period- 55 month median
Measure: Number; unit: participants
Arm/Group | EDTA + High Dose Vitamin | EDTA + High Dose Vitamin Placebo | EDTA Placebo + High Dose Vitamin | EDTA Placebo + High Dose Vitamin Placebo
Number analyzed (Participants) | 421 | 418 | 432 | 437
participants | 108 | 114 | 122 | 139

2. Secondary Outcome: A Composite of Cardiovascular Death, Non-fatal Myocardial Infarction and Non-fatal Stroke.
Description: Number of patients with events (composite of cardiovascular death, non-fatal MI, non-fatal stroke) Events were centrally adjudicated where available; otherwise site reported events were used.
Time Frame: Measured over a maximum 5-year follow-up period- 55 month median
Measure: Number; unit: participants
Arm/Group | EDTA + High Dose Vitamin | EDTA + High Dose Vitamin Placebo | EDTA Placebo + High Dose Vitamin | EDTA Placebo + High Dose Vitamin Placebo
Number analyzed (Participants) | 421 | 418 | 432 | 437
participants | 39 | 57 | 55 | 58

ADVERSE EVENTS:
Arm/Group | EDTA + High Dose Vitamin | EDTA + High Dose Vitamin Placebo | EDTA Placebo + High Dose Vitamin | EDTA Placebo + High Dose Vitamin Placebo
Serious Adverse Events (participants affected / at risk) | 2/421 | 0/418 | 0/432 | 2/437
Other Adverse Events (participants affected / at risk) | 168/421 | 201/418 | 164/432 | 185/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDTA + High Dose Vitamin (N=421) | EDTA + High Dose Vitamin Placebo (N=418) | EDTA Placebo + High Dose Vitamin (N=432) | EDTA Placebo + High Dose Vitamin Placebo (N=437)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EDTA + High Dose Vitamin (N=421) | EDTA + High Dose Vitamin Placebo (N=418) | EDTA Placebo + High Dose Vitamin (N=432) | EDTA Placebo + High Dose Vitamin Placebo (N=437)
Diarrhoea (Gastrointestinal disorders) | 15 | 16 | 23 | 23
Nausea (Gastrointestinal disorders) | 17 | 22 | 16 | 19
White Blood Cell Count Decreased (Investigations) | 13 | 27 | 16 | 19
Hypocalcaemia (Metabolism and nutrition disorders) | 63 | 69 | 34 | 43
Hypoglycaemia (Metabolism and nutrition disorders) | 40 | 48 | 49 | 54
Proteinuria (Renal and urinary disorders) | 20 | 19 | 26 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Enrolling Centers must abide by all TACT and NIH conflict of interest policies. Decisions about authorship on all multi-center publications resulting from research under this agreement will be made by the TACT Publica¬tions Committee prior to publication. No publications or other public disclosure shall be made until the TACT results are unblinded and results from all sites have been received and analyzed or TACT has been abandoned at all sites.